CLINICAL TRIAL: NCT01874028
Title: A Phase 1 Pharmacokinetic Profiling Study in Patients Receiving Trientine Dihydrochloride for the Treatment of Wilson's Disease.
Brief Title: A Phase 1 Study to Assess the Effects in the Body of a Single Dose of Trientine Dihydrochloride in Wilson's Disease Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Univar BV (Industry)
Collaborators: Aptiv Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TR-001PK
Record Dates: First submitted 2013-06-06; First posted 2013-06-10 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Wilson's Disease
Keywords: Trientine; Pharmacokinetics
MeSH Terms: conditions — Hepatolenticular Degeneration | interventions — Trientine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trientine dihydrochloride (Experimental)
  Interventions: Drug: trientine dihydrochloride

INTERVENTIONS:
Drug: trientine dihydrochloride — Patients will take their normal prescribed dose (x1) of trientine dihydrochloride 300mg

SUMMARY:
To evaluate the effects of a single dose of trientine in children ≥6 years and adult patients with Wilson's disease.

DETAILED DESCRIPTION:
An open, single-dose study to determine the pharmacokinetics, and safety of oral administration of trientine dihydrochloride in both children and adult patients with Wilson's Disease. Blood samples will be taken pre-dose and at 10 time-points post-dose to investigate the pharmacokinetic profile of trientine dihydrochloride up to 12 hours after intake of study medication in 20 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Children ≥ 6 years and adult patients
2. Confirmed diagnosis of Wilson's disease by Leipzig-Score >3 (Ferenci et al 2003)
3. Current treatment with trientine dihydrochloride
4. Signed informed consent including parental consent in patients ≤ 18 years
5. Agree to remain in the study site1 for the PK measurements period.

Exclusion Criteria:

1. Known clinically significant allergy or hypersensitivity to drugs that, in the opinion of the investigator, may affect the patient's safety
2. Have any clinically significant conditions that would interfere with the collection or interpretation of the study results or would compromise the patient's health
3. Women of child bearing potential who do not use contraceptives, breastfeeding, or pregnant women
4. Severe anaemia (haemoglobin <9 mg/dL)
5. In the judgment of the Investigator, is likely to be noncompliant or uncooperative during the study, or unable to cooperate because of a language problem or poor mental development
6. Participation in any interventional clinical study at the same time or within the 4 weeks prior his study.

Ages: 6 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic measurements | Evaluation of PK parameters will occur at 11 time points:Pre-dose), and at 30 minutes, 1, 1.5, 2, 3, 4, 5, 6, 8, and 12 hours post-dose
  The main objective of the study is to evaluate the pharmacokinetics of a single dose of trientine dihydrochloride in children ≥6 years and adult patients with Wilson's disease by PK analysis.
  Non-compartmental or model-independent methods will be used to derive pharmacokinetic parameters using individual patient plasma concentration-time data. Pharmacokinetic parameters will include the Cmax, Tmax, T1/2, and the concentration-time curved (AUC0-t) and AUCinf.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinik Heidelberg, Heidelberg, Germany